CLINICAL TRIAL: NCT03811756
Title: The Effect of 12-week Dietary Intake of Syrup Containing CoQ10 and Collagen on Dermis Density and Other Skin Parameters: Randomised Double-blind Placebo-controlled Study
Brief Title: The Effect of 12-week Dietary Intake of Syrup Containing CoQ10 and Collagen on Dermis Density and Other Skin Parameters
Acronym: Q10-collagen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: European Regional Development Fund (Other); Valens Int. d.o.o., Slovenija (Industry); Ministry of Education, Science and Sport, Republic of Slovenia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIST F4F Q10-collagen 01-2018
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2019-12

CONDITIONS: Dermis Density; Trans Epidermal Water Loss (TEWL); Skin Hydration; Wrinkles; Dermis Thickness
MeSH Terms: interventions — Collagen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator): Participants will receive investigational product - Test syrup containing CoQ10 and collagen (daily dose 10 mL: fish collagen (Peptan®): 4000 mg, water soluble CoQ10 (Q10Vital®): 50 mg, vitamin C: 80 mg, vitamin A: 920 μg, biotin: 150 μg).
  Interventions: Dietary Supplement: Test syrup containing CoQ10 and collagen
- Placebo group (Placebo Comparator): Placebo group participants will receive placebo syrup without active ingredients. (daily dose 10 mL: fish collagen: 0 mg, water soluble CoQ10 (Q10Vital®): 0 mg, vitamin C: 0 mg, vitamin A: 0 μg, biotin: 0 μg); continous administration of placebo product for 12 weeks.
  Interventions: Dietary Supplement: Placebo syrup

INTERVENTIONS:
Dietary Supplement: Test syrup containing CoQ10 and collagen — Test group will receive investigational product - test syrup (daily dose 10 mL: fish collagen: 4000 mg, water soluble CoQ10 (Q10Vital®): 50 mg, vitamin C: 80 mg, vitamin A: 920 μg, biotin: 150 μg); continuous administration of investigational product for 12 weeks.
  Arms: Test group
Dietary Supplement: Placebo syrup — Placebo group will receive placebo syrup without active ingredients. (daily dose 10 mL: fish collagen: 0 mg, water soluble CoQ10 (Q10Vital®): 0 mg, vitamin C: 0 mg, vitamin A: 0 μg, biotin: 0 μg); continous administration of placebo product for 12 weeks.
  Arms: Placebo group

SUMMARY:
Placebo controlled double-blind multi-dose comparative study of the effects of coenzyme Q10 and collagen formulation with improved water-solubility in healthy adults.

One group (test group) will receive investigational product - test syrup (daily dose 10 mL: fish collagen: 4000 mg, water soluble CoQ10 (Q10Vital®): 50 mg, vitamin C: 80 mg, vitamin A: 920 μg, biotin: 150 μg) and the other (placebo group) placebo syrup without those active ingredients. Participants will test continuous administration of placebo or investigational product for 12 weeks in order to demonstrate and assess multiple-dose effects on skin condition and signs of skin aging.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian female volunteers aged between 40 and 65 years at the time of the signature of Informed consent form (ICF),
* Signed Informed consent form (ICF),
* Fitzpatrick skin phototypes II and III,
* Signs of skin aging,
* In good health condition,
* Willingness to avoid a consumption of any food supplements containing CoQ10 and other antioxidants, collagen or vitamins during the study,
* Willingness to follow all study procedures and keeping a diary during the study (to follow their compliance and palatability).

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Known or suspected allergy to any ingredient of the tested products,
* Changes in dietary habits and dietary supplementation in last three months prior to inclusion,
* Regular use of food supplements containing CoQ10 or other antioxidants, collagen or other protein-based food supplements, vitamin A, vitamin E or biotin in last three months prior to inclusion,
* Veganism,
* Changes in cosmetic facial and body care routine in last month prior to inclusion,
* Diagnosed and uncontrolled/untreated/unregulated disease,
* Any clinically significant history of serious metabolic disease, digestive tract disease, liver disease, kidney disease, haematological disease,
* Acute skin diseases,
* Skin pigmentation disorders,
* Increased cholesterol and use of cholesterol lowering drugs (statins),
* Anticipated sunbathing or solarium visits before or during the study,
* Invasive rejuvenation treatments (e.g. needle rollers, needle mesotherapy, deep/medium-deep chemical peels etc.) in last 6 months prior to study entry,
* Non-invasive rejuvenation treatments (e.g. radiofrequency, electrotherapy, ultrasound therapy) in last 2 months prior to study entry,
* Mental incapacity that precludes adequate understanding or cooperation.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Influence of investigational product in relation to placebo product on dermis density assessed through dermis intensity measurement | 12 weeks
  Significant change of dermis density from baseline in test group, in comparison to placebo group after 12 weeks of dietary supplementation with study product is expected. Dermis density will be assessed through ultrasonographic dermis intensity measurement.

SECONDARY OUTCOMES:
Influence of the investigational product in relation to placebo product on skin elasticity assessed through measurements of viscoelasticity | 12 weeks
  For assessments of skin viscoelasticity measurements will be performed. Significant change of skin viscoeasticity from baseline in test group, in comparison to placebo group after 12 weeks of dietary supplementation with study product is expected.
Influence of the investigational product in relation to placebo product on skin hydration | 12 weeks
  Assessment of the effects of the investigational product on skin hydration after 12 weeks of dietary supplementation. Skin hydration measurements will be performed using conductance principle.
Influence of the investigational product in relation to placebo product on TEWL | 12 weeks
  Assessment of the effects of investigational product on transepidermal water loss after 12 weeks of dietary supplementation. TEWL measurements will be performed using open chambre principle.
Influence of investigational product in relation to placebo product on dermis thickness | 12 weeks
  Significant change of dermis thickness from baseline in test group, in comparison to placebo group after 12 weeks of dietary supplementation with study product is expected. Dermis density will be assessed using ultrasonography.
Influence of investigational product in relation to placebo product on wrinkles will be assessed using wrinkle area fraction measurements | 12 weeks
  Assessment of the effects of investigational product on facial wrinkles after 12 weeks of dietary supplementation will be done using wrinkle area fraction measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Study Director — Head of Reasearch Group
Locations (1):
- Higher School of Applied Sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No